CLINICAL TRIAL: NCT05732779
Title: Mobile Video Directly Observed Therapy (DOT) for Immunosuppression Medication Adherence in Adolescent Heart Transplant Recipients: Enhancing Technological Innovation and Strengthening the Role of Small Businesses in Meeting Needs of Adolescent Organ Transplant
Brief Title: Mobile Video Directly Observed Therapy (DOT) for Immunosuppression Medication Adherence in Adolescent Heart Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: emocha Mobile Health, Inc. (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201809; R44HL167591-01A1 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Heart Transplant Rejection; Immune Suppression; Pediatric Heart Transplant; Medication Nonadherence; Health Behavior; Remote Monitoring; Patient Engagement
MeSH Terms: conditions — Medication Adherence; Health Behavior; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eMocha intervention (Experimental): Adolescent patients randomized to the use of asynchronous mobile video directly observed therapy (DOT) intervention (eMocha DOT app)
  Interventions: Other: DOT intervention
- Standard of care (No Intervention): Adolescent patients who continue enhanced goal-setting standard of care

INTERVENTIONS:
Other: DOT intervention — A mobile health application developed by eMocha Health Inc. facilitates asynchronous mobile video directly observed therapy (DOT) intervention, empowering users to track dose-by-dose medication adherence
  Arms: eMocha intervention

SUMMARY:
We will conduct a two-group randomized controlled trial to examine the eMocha DOT intervention with pediatric HT recipients.In this population, medication nonadherence remains a primary cause of late acute rejection (LAR) episodes, increased number of hospitalizations, graft failure, and patient mortality. Herein, we propose an innovative approach to promote medication adherence and improve patient and graft outcomes.

DETAILED DESCRIPTION:
Few interventions have proven to be successful in promoting medication adherence and impacting short- and long-term post-transplant outcomes in adolescent heart transplant (HT) recipients. Improving adherence is a persistent challenge with youth experiencing chronic health conditions, especially among adolescent transplant recipients. Adolescent organ transplant recipients experience unique challenges remaining adherent to the complex post-transplant regimen, with rates of non-adherence as high as 40% to 60%. In this population, medication non-adherence remains a primary cause of late acute rejection (LAR) episodes, increased number of hospitalizations, graft failure, and patient mortality. Herein, we propose an innovative approach to promote medication adherence and improve patient and graft outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are 10-21 years of age
* Have received a heart transplant and are followed participating pediatric heart transplant centers
* English-speaking or Spanish-speaking
* Own a smart-phone or have access to the mobile app through other devices
* Are willing to receive information through it
* Have a MLVI score of greater than 2.0 over the last year

Exclusion Criteria:

• Those with cognitive impairments will not be eligible for enrollment due to inability to provide informed assent

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence based on medication level variability index | 12 weeks
  medication level variability index (MLVI). MLVI is calculated as the Standard Deviation of a set of at least 3 tacrolimus trough blood levels for each participant.
Directly observed medication adherence | 1 weeks
  Number of doses observed and reviewed by nursing staff compare to number of prescribed doses per day
Late Acute Rejection | 6 months post-intervention
  Number of biopsy-proven rejection, clinician-assigned rejection
Hospitalization | 6 months post-intervention
  Number of hospitalizations
Patient Activation Measure | Pretest at enrollment and posttest at 12 weeks
  A 13-item scale designed to measure a patient's perception of their knowledge, skill and confidence in managing their chronic health condition
Patient Assessment of Chronic Illness Care (PACIC) | Pretest at enrollment and posttest at 12 weeks
  A 20-item scale with five subscales (scale of 1 (none) to 5 (always), total score 20 to 200, higher score being better outcome) that assess patient activation, delivery system design, goal setting, problem-solving and contextual counseling, and follow-up and coordination.
Self-reported user satisfaction with the DOT app | Pretest at enrollment and posttest at 12 weeks
  Collected using a modified version of the engagement index questionnaire used
Engagement metrics | Pretest at enrollment and posttest at 12 weeks
  Standard engagement metrics or paradata (e.g., amount, frequency, duration, and depth of use)
PedsQL 3.0 Transplant Module (PedsQL-TM) | Pretest at enrollment and posttest at 12 weeks
  HRQOL
Adolescent Medication Barriers Scale (AMBS) | Pretest, posttest
  To assess adolescent perceived barriers to medication adherence
Parent Medication Barriers Scale (PMBS) | Pretest at enrollment and posttest at 12 weeks
  To assess parental perceived barriers to their child taking their medication

CONTACTS AND LOCATIONS:
Overall Officials: Dipankar Gupta, MD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - University of Miami, Miller School of Medicine, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - FSU College of Medicine, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No